CLINICAL TRIAL: NCT03647839
Title: Modulation Of The Tumour Microenvironment Using Either Vascular Disrupting Agents or STAT3 Inhibition in Order to Synergise With PD1 Inhibition in Microsatellite Stable, Refractory Colorectal Cancer
Acronym: MODULATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-99U
Record Dates: First submitted 2018-07-02; First posted 2018-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Microsatellite stable tumour; Refractory colorectal cancer; Tumour microenvironment; Vascular Disrupting Agent; STAT3 inhibitors; PD1 inhibitors; Unresectable colorectal cancer; nivolumab; BNC105; BBI-608
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab; BNC 105; napabucasin

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicentre, parallel phase II study designed to assess the efficacy of the combination of nivolumab and BNC105 and the combination of nivolumab and BBI-608. Patients with microsatellite stable adenocarcinoma of colorectal origin that is not resectable are eligible and will be randomised in the ratio of 1:1 using permuted block randomisation with stratification by screening ECOG performance status (0 or 1) to receive either nivolumab and BNC105 or nivolumab and BBI-608.
Masking Description: This is an open-label, multicentre, parallel phase II study designed to assess the efficacy of the combination of nivolumab and BNC105 and the combination of nivolumab and BBI-608. Patients with microsatellite stable adenocarcinoma of colorectal origin that is not resectable are eligible and will be randomised in the ratio of 1:1 using permuted block randomisation with stratification by screening ECOG performance status (0 or 1) to receive either nivolumab and BNC105 or nivolumab and BBI-608.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 (Experimental): Nivolumab and BNC105
  Interventions: Drug: Nivolumab 10 MG/ML; Drug: BNC 105
- Arm 2 (Experimental): Nivolumab and BBI-608
  Interventions: Drug: Nivolumab 10 MG/ML; Drug: BBI608

INTERVENTIONS:
Drug: Nivolumab 10 MG/ML — Nivolumab will be supplied free of charge by Bristol-Myers Squibb (BMS) as sterile liquid in 10mL glass vials.
  Other Names: Opdivo
Drug: BNC 105 — BNC105 will be provided free of charge by Bionomics, as a sterile solution of BNC105P. BNC105P is a clear, colorless to yellow liquid presented in a clear glass vial and is intended to be diluted with commercially available sterile 0.9% saline prior to IV administration.
  Arms: Arm 1
Drug: BBI608 — BBI-608 will be supplied free of charge by Boston Biomedical as capsules.
  Other Names: Napabucasin
  Arms: Arm 2

SUMMARY:
This Phase II research project will test the efficacy, safety, and tolerability of an experimental drug combination: either nivolumab and BBI608 or nivolumab and BNC105 in patients with metastatic colorectal cancer who have previously failed standard of care treatment.

DETAILED DESCRIPTION:
This is an open-label, multicentre, parallel phase II study designed to assess the efficacy of the combination of nivolumab and BNC105 and the combination of nivolumab and BBI-608. Patients with microsatellite stable adenocarcinoma of colorectal origin that is not resectable are eligible and will be randomised in the ratio of 1:1 using permuted block randomisation with stratification by screening ECOG performance status (0 or 1) to receive either nivolumab and BNC105 or nivolumab and BBI-608.

The expected sample size is 90 patients over a 24 month recruitment period.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a histological diagnosis of adenocarcinoma of colorectal origin.
2. Has documented microsatellite stable tumour as assessed by PCR or IHC.
3. Metastatic disease that is not resectable.
4. Male or female patients > 18 years of age at screening.
5. Failed in any sequence or combination oxaliplatin, fluoropyrimidine, irinotecan with or without bevacizumab where failure is defined as progression or toxicity precluding further therapy.
6. For patients with ras/b-raf wild type tumours: failed anti EGFR therapy (cetuximab and/or panitumumab) where failure is defined as progression or toxicity precluding further therapy. Patients with b-raf mutant tumours and/or right sided primary tumours may have received anti-EGFR therapy but this is not mandated.
7. Patient has measurable disease according to RECIST 1.1.
8. Metastatic lesion(s) amenable to biopsy, this cannot be the sole site of measurable disease.
9. ECOG performance status 0 or 1.
10. Adequate organ and hematologic function within 7 days of randomisation, defined by:

    1. Neutrophils > 1.5 X 109/L
    2. Platelets > 80 X 109/L
    3. Serum aspartate transaminase (AST) or alanine transaminase (ALT) < 3 x upper limit of normal (ULN)
    4. Bilirubin < 1.5 x ULN
    5. Albumin >30g/L
    6. Creatinine clearance ≥ 50ml/min(Cockcroft-Gault).
11. Life expectancy of at least 12 weeks
12. No other concurrent uncontrolled medical conditions
13. No other malignant disease apart from non-melanotic skin cancer or carcinoma in situ of the uterine cervix or any other cancer treated with curative intent >2 years previously without evidence of relapse.
14. Female patients of childbearing potential should have a negative urine or serum pregnancy within 24 hours prior to randomisation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
15. Female patients of childbearing potential should be willing to use a reliable method of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 180 days after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
16. Male patients with female partners of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy.
17. Patient has provided written informed consent including consent for tumour biopsies and donation of tumour tissue for biomarker studies.

Exclusion Criteria:

1. Medical or psychiatric conditions that compromise the patient's ability to give informed consent or to complete the protocol.
2. Patients with any active, known, or suspected autoimmune disease, with the following exceptions:

   1. Patients with vitiligo, type 1 diabetes mellitus, resolved childhood asthma or atopy are permitted to enroll.
   2. Patients with suspected autoimmune thyroid disorders may be enrolled if they are currently euthyroid or with residual hypothyroidism requiring only hormone replacement.
   3. Patients with psoriasis requiring systemic therapy must be excluded from enrolment
3. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg/day prednisone equivalent) or other immunosuppressive medications within 14 days of randomisation. Inhaled or topical steroids and adrenal replacement doses > 10mg/day prednisone equivalents are permitted in the absence of active autoimmune disease.
4. Patient has evidence of interstitial lung disease or active, non-infectious pneumonitis.
5. Has an active infection requiring systemic therapy.
6. Patients receiving long-term anti-coagulation or anti-platelet agents which cannot be ceased for an appropriate interval to allow mandatory tumour biopsies prior to and during therapy.
7. Patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate.
8. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
9. Has a known history of HIV (HIV 1/2 antibodies). Formal testing is only required if there is significant clinical suspicion of HIV.
10. Known active brain metastases (unless adequately treated with surgery and/or radiotherapy >30 d prior and asymptomatic).
11. Significant vascular events within the previous 6 months (unstable angina, myocardial infarction, TIA, CVA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Objective response per iRECIST | From start of treatment up to the date when the last patient has their 6 months follow-up assessment

SECONDARY OUTCOMES:
Objective response per RECIST1.1 | From start of treatment up to the date when the last patient has their 6 months follow-up assessment
Progression free survival (PFS). | From start of treatment until the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to the date when the last patient has their 6 months follow-up assessment
Adverse event assessed using CTCAE version 5.0 | Through treatment completion, maximum of 2 years
Overall survival | From start of treatment until the date of death from any cause, assessed up to the date when the last patient has their 6 months follow-up assessment

CONTACTS AND LOCATIONS:
Overall Officials: Niall Tebbutt, Prof, Study Chair — Olivia Newton-John Cancer Wellness and Research Centre
Locations (14):
- Australia (14):
  - Border Cancer Hospital, Albury, New South Wales
  - Newcastle Private Hospital, Newcastle, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Queen Elizabeth Hospital, Woodville South, South Australia
  - Ballarat Health Service, Ballarat, Victoria
  - Eastern Health, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - Olivia Newton-John Cancer Wellness and Research Centre, Heidelberg, Victoria
  - Peninsula Health/Frankston Hospital, Mornington Peninsula, Victoria
  - Western Health, Saint Albans, Victoria

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.